CLINICAL TRIAL: NCT02996305
Title: A Phase 2 Adult and Adolescent Angelman Syndrome Clinical Trial: A Randomized, Double-Blind, Safety and Efficacy Study of Gaboxadol
Brief Title: A Study in Adults and Adolescents With Angelman Syndrome (STARS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OV101-15-001
Record Dates: First submitted 2016-12-02; First posted 2016-12-19 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome | interventions — gaboxadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OV101 regimen 1 (Experimental): OV101 once daily
  Interventions: Drug: OV101 Regimen 1
- OV101 regimen 2 (Experimental): OV101 twice daily
  Interventions: Drug: OV101 regimen 2
- Placebo (Placebo Comparator): Twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: OV101 Regimen 1
  Other Names: Gaboxadol
  Arms: OV101 regimen 1
Drug: OV101 regimen 2
  Other Names: Gaboxadol
  Arms: OV101 regimen 2
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety and tolerability of oral OV101 (gaboxadol) in adult and adolescent subjects with Angelman syndrome. In addition, several exploratory efficacy outcome measures will be investigated.

DETAILED DESCRIPTION:
Two dosing schedules of OV101 (gaboxadol) giving as once daily or twice daily dose will be assessed against placebo.

ELIGIBILITY:
Inclusion Criteria

1. Age 13- 49 years
2. Diagnosis of Angelman syndrome
3. Receiving a stable regimen of concomitant medications for at least 4 weeks prior to Baseline, and able to maintain these throughout the duration of the study
4. Has a caregiver capable of providing informed consent on behalf of the subject and able to attend scheduled study visits
5. Able to ingest study medication
6. Caregivers must agree not to post any subject or study information on social media

Exclusion Criteria

1. Unable to perform the study related safety and exploratory efficacy assessments, such as motor function
2. Poorly controlled seizure activity
3. Concomitant cardiovascular, respiratory, liver, renal, or hematologic diseases of a degree that would limit participation in the study
4. Pregnancy or women of child-bearing potential who are not using and acceptable method of contraception
5. Concomitant use of minocycline, levodopa, zolpidem, zaleplon, eszopiclone, ramelteon, and cannabinoid derivatives, or any other use of any investigational agent, device, and/or investigational procedure 4 weeks prior to Baseline and during the study
6. Allergy to OV101 or any excipients
7. At increased risk of harming self and/or others based on investigator assessment
8. Any condition or reason that in the opinion of the investigator makes the subject unsuitable for enrollment
9. Inability of subject or caregiver to comply with study requirements

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 13 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06-07 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Rakhit, MD, MBA, Study Director — Healx AI
Locations (13):
- United States (12):
  - Ovid Therapeutics Investigative Site, Phoenix, Arizona
  - Ovid Therapeutics Investigative Site, San Diego, California
  - Ovid Therapeutics Investigative Site, Gainesville, Florida
  - Ovid Therapeutics Investigative Site, Tampa, Florida
  - Ovid Therapeutics Investigative Site, Atlanta, Georgia
  - Ovid Therapeutics Investigative Site, Chicago, Illinois
  - Ovid Therapeutics Investigative Site, Boston, Massachusetts
  - Ovid Therapeutics Investigative Site, Lexington, Massachusetts
  - Ovid Therapeutics Investigative Site, Cincinnati, Ohio
  - Ovid Therapeutics Investigative Site, Media, Pennsylvania
  - Ovid Therapeutics Investigative Site, Greenwood, South Carolina
  - Ovid Therapeutics Investigative Site, Nashville, Tennessee
- Ovid Therapeutics Investigative Site, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bird LM, Ochoa-Lubinoff C, Tan WH, Heimer G, Melmed RD, Rakhit A, Visootsak J, During MJ, Holcroft C, Burdine RD, Kolevzon A, Thibert RL. The STARS Phase 2 Study: A Randomized Controlled Trial of Gaboxadol in Angelman Syndrome. Neurology. 2021 Feb 16;96(7):e1024-e1035. doi: 10.1212/WNL.0000000000011409. Epub 2020 Dec 21. PMID 33443117

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Giving twice daily
- OV101 QD: OV101, once daily (15mg night)
- OV101 BID: OV101, twice daily (10mg morning, 15mg night)
Period: Overall Study
Arm/Group | Placebo | OV101 QD | OV101 BID
Started | 29 | 29 | 30
Completed | 26 | 27 | 25
Not Completed | 3 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo BID Evening and Morning
- OV101 QD: OV101 15 mg Evening Placebo in the Morning
- OV101 BID: OV101 15 mg Evening OV101 10 mg Morning
- Total: Total of all reporting groups
Arm/Group | Placebo | OV101 QD | OV101 BID | Total
Number analyzed (Participants) | 29 | 29 | 29 | 87
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at Inform Consent | 22.0 (6.70) | 23.1 (7.76) | 22.8 (6.51) | 22.6 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 11 | 34
  Male | 15 | 20 | 18 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 5 | 14
  Not Hispanic or Latino | 26 | 23 | 23 | 72
  Unknown or Not Reported | 0 | 0 | 1 | 1
Gender [Count of Participants; unit: Participants]
  Male | 15 | 20 | 18 | 53
  Famale | 14 | 9 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events in Placebo and Active Treatment Groups
Description: Summary of Subjects Reporting at least one Treatment Emergent Adverse Event (TEAEs), Safety Set. The table below summarizes the subjects who experienced TEAEs in the study.
Time Frame: Baseline and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OV101 QD | OV101 BID
Number analyzed (Participants) | 29 | 29 | 29
Participants
  Any TEAE | 25 | 27 | 25
  Any Mild TEAE | 23 | 23 | 23
  Any Moderate TEAE | 9 | 15 | 9
  Any Severe TEAE | 0 | 1 | 4
  Any Life-Threatening TEAE | 0 | 0 | 0
  Drug-related TEAE | 13 | 18 | 19
  Any Serious TEAE | 0 | 1 | 1
  Any TEAE leading to Dose Change or Interruption | 5 | 5 | 8
  Any TEAE Leading to Study Withdrawal | 1 | 0 | 3

2. Primary Outcome: Incidence of Adverse Events in Placebo and Active Treatment Groups
Description: The Treatment Emergent Adverse Event (TEAEs) Reported by ≥10% of Subjects in Any Treatment Group by Preferred Term, Safety Set.
Time Frame: Baseline and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OV101 QD | OV101 BID
Number analyzed (Participants) | 29 | 29 | 29
Participants
  At least 1 TEAE | 25 | 27 | 25
  Vomiting | 9 | 5 | 5
  Somnolence | 5 | 5 | 3
  Irritability | 4 | 3 | 5
  Pyrexia | 2 | 7 | 1
  Upper respiratory tract infection | 4 | 5 | 1
  Aggression | 5 | 4 | 1
  Rash | 1 | 3 | 2
  Seizure | 0 | 2 | 3
  Decreased appetite | 4 | 2 | 2
  Diarrhoea | 3 | 1 | 3
  Nausea | 3 | 0 | 4
  Nasopharyngitis | 5 | 2 | 1

3. Primary Outcome: Incidence of Adverse Events in Placebo and Active Treatment Groups
Description: Treatment-related TEAEs (Treatment Emergent Adverse Event) in ≥ 2 Subjects in OV101 Combined, Safety Set. The incidence of TEAEs assessed as treatment-related (at least possibly related to study drug, by the Investigator). Preferred Term in the table below.
Time Frame: Baseline and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OV101 QD | OV101 BID
Number analyzed (Participants) | 29 | 29 | 29
Participants
  At least 1 Treatment-related TEAE | 13 | 18 | 19
  Nausea | 2 | 0 | 2
  Fatigue | 2 | 1 | 2
  Decreased appetite | 2 | 0 | 2
  Somnolence | 5 | 5 | 2
  Myoclonic epilepsy | 0 | 1 | 2
  Myoclonus | 0 | 1 | 2
  Seizure | 0 | 1 | 2
  Lethargy | 0 | 0 | 2
  Sedation | 0 | 1 | 1
  Tremor | 0 | 1 | 1
  Irritability | 3 | 2 | 4
  Aggression | 2 | 4 | 1
  Insomnia | 1 | 2 | 1
  Agitation | 0 | 1 | 2
  Anxiety | 0 | 0 | 2
  Enuresis | 0 | 1 | 1
  Sleep disorder | 0 | 0 | 2
  Rash | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: 12 Weeks
Groups:
- Placebo: Placebo Morning and Evening
- OV101 QD: OV101 15mg Evening
Arm/Group | Placebo | OV101 QD | OV101 BID
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/29 | 1/29
Other Adverse Events (participants affected / at risk) | 13/29 | 18/29 | 19/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | OV101 QD (N=29) | OV101 BID (N=29)
Seizure (Nervous system disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | OV101 QD (N=29) | OV101 BID (N=29)
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
General disorders and administration site conditions (Nervous system disorders) | 5 | 3 | 2
Fatigue (General disorders) | 2 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2
Somnolence (Nervous system disorders) | 5 | 5 | 2
Myoclonus (Nervous system disorders) | 0 | 1 | 2
Seizure (Nervous system disorders) | 0 | 1 | 2 — Seizures include both Seizures and Myclonic jerks, both of which were balanced across all treatment groups.
Lethargy (Nervous system disorders) | 0 | 0 | 2
Irritability (Psychiatric disorders) | 3 | 2 | 4
Aggression (Psychiatric disorders) | 2 | 4 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Myoclonic epilepsy (Nervous system disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication

1. Institution/Investigator will submit to Sponsor any paper relating to the Study 60 days prior to disclosure. If Sponsor wants a patent to be filed on Inventions, then the period shall be extended by 90 days
2. Multi-center Studies.Institution/Investigator may publish a paper in its performance of Study after the later of (a) publication of the multi-center publication; (b) confirmation there will be no multi-center publication; or(c) 36 months after the completion of the Study

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT02996305/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan document (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02996305/SAP_001.pdf